CLINICAL TRIAL: NCT05144087
Title: The Influence of Mepolizumab on Structural and Inflammatory Cells in Severe Eosinophilic Asthma
Acronym: IRIS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM MED1765
Record Dates: First submitted 2021-09-03; First posted 2021-12-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Asthma; Eosinophilic
Keywords: asthma; mepolizumab; eosinophil
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bronchial epithelial cells bronchoalveolar lavage (BAL) peripheral airway brushings blood serum and plasma urinary metabolites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The IRIS study aims to investigate the way Mepolizumab affects the structure of the airway cells in patients with Severe Eosinophilic Asthma and how the immune function of these cells changes with treatment. The aim is to take samples of cells from the airways before starting Mepolizumab and after 6 months of treatment. These samples will be taken during a bronchoscopy (a camera test looking into the lungs) and we will analyse these cells in the laboratory. These investigations will allow us to better understand how Mepolizumab affects the cells within the airways.

DETAILED DESCRIPTION:
IRIS is a prospective observational study investigating Mepolizumab in the treatment of severe eosinophilic asthma.

Eosinophilic airway inflammation has been implicated in the pathogenesis of asthma and is particularly relevant in severe eosinophilic asthma (SEA), in which standard asthma therapies fail to adequately control the disease. In severe asthma, there is bronchial epithelial damage and loss of tight junction integrity, goblet cell hyperplasia, enhanced collagen generation within the airway wall and impaired innate immune responses. Mepolizumab has been shown to reduce exacerbations and improve disease control in SEA but there are no studies assessing the impact of Mepolizumab on structural airway cell activity and function and airway remodelling processes.

Primary Objective:

To investigate changes within bronchial epithelial cells following completion of 6 months (7 doses) of Mepolizumab using single cell RNA sequencing (scRNA-seq) and Frac-seq (subcellular fractionation and RNA-sequencing).

Secondary Objectives:

To investigate the following after completing treatment with 6 months of Mepolizumab:

i) Changes in epithelial barrier integrity using Frac-seq, transepithelial resistance ii) Changes in epithelial antiviral responses fusing Frac-seq in unstimulated and virus-infected cells.

iii) Changes in airway remodelling by assessing the profile of fibroblasts isolated from bronchial biopsies employing Frac-seq and immunostaining of bronchial biopsies iv) Evaluate the impact on peripheral airways by obtaining bronchoalveolar lavage (BAL) and peripheral airway brushings for Frac-seq analysis and protein analysis v) Peripheral airway dysfunction using impulse oscillometry vi) Changes in fibroblast profile with stimulation and IL-5 inhibition using a range of molecular, cellular, protein and metabolic techniques

Exploratory Objectives i) Evaluation of neural structural changes using biopsies

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Severe Eosinophilic Asthma (as per Southampton Severe Asthma MDT and based on ATS/ERS consensus criteria)
2. Approved for treatment with Mepolizumab by Southampton Severe Asthma MDT (in accordance with NICE TA 431)

   * Blood eosinophil count is ≥0.3 x109cells/L in preceding 12 months
   * ≥4 asthma exacerbations needing systemic steroids in the preceding 12 months
3. Age ≥18 years
4. Able to provide written informed consent

Exclusion Criteria:

1. On maintenance daily oral steroids, asthma immune modulators
2. On long-term systemic antibiotics or antifungal treatment
3. Current smoker or ex-smoker with >10 pack year smoking history
4. Known clinically significant respiratory disorder such as bronchiectasis, interstitial lung disease, allergic bronchopulmonary aspergillosis
5. Currently pregnant or planning pregnancy within the treatment period or breast-feeding
6. History of psychiatric, medical or surgical disorders that in the opinion of the chief investigator may interfere with undergoing a bronchoscopy or may compromise study completion or data collection
7. Current malignancy
8. Alcohol or recreational drug abuse
9. Diagnosis of immunodeficiency requiring treatment
10. Previous bronchial thermoplasty
11. Previous treatment with biological therapy
12. Previously unable to tolerate a bronchoscopy
13. Current or recent (within the last 12 weeks) infection with SARS-CoV-2
14. Unable to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from University Hospital Southampton (UHS). UHS operates a regional specialist clinical severe asthma service, prescribing biological therapies, including Mepolizumab. Patients will be exclusively recruited from a pool of patients awaiting biological therapies for severe asthma at these centres. Patients are only eligible for Mepolizumab following NICE mandated multidisciplinary team approval reviewing biological eligibility, treatment adherence and satisfaction that other co-morbid conditions have been satisfactorily addressed.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
To investigate molecular changes in the bronchial epithelium that occurs with mepolizumab treatment using RNA sequencing | 36 months
  Changes at the level of single cell RNA sequencing will be reported as:
  1. Changes in the percentage of cell populations present in the airways
  2. Normalised gene counts

SECONDARY OUTCOMES:
Changes in epithelial barrier integrity using transepithelial resistance | 36 months
  Transepithelial resistance measures changes in voltage across the epithelial cells
Changes in epithelial antiviral responses using interferon and other antiviral gene measurements | 36 months
  Gene expression will be measured using RNA sequencing and reported as gene counts
Changes in airway remodelling by assessing fibroblasts isolated from bronchial biopsies using RNA sequencing | 36 months
  RNA sequencing will be reported as gene counts
Changes in airway remodelling by assessing fibroblasts isolated from bronchial biopsies using immunostaining | 36 months
  Immunostaining will be reported as mean fluorescence intensity and percentage of cells stained
Evaluate the impact of Mepolizumab on peripheral airways by obtaining bronchoalveolar lavage for RNA sequencing | 36 months
  RNA sequencing will be reported as gene counts
Evaluate the impact on peripheral airways by obtaining peripheral airway brushings for RNA sequencing | 36 months
  RNA sequencing will be reported as gene counts
Peripheral airway dysfunction using impulse oscillometry | 36 months
  Impulse oscillometry will be measured as resistance and impedance
Changes in fibroblast profile with stimulation and IL-5 inhibition using a range of molecular, cellular, protein and metabolic techniques | 24 Months
  To study fibroblasts

OTHER OUTCOMES:
Evaluation of neural structural changes using immunostaining on biopsy specimens | 36 months
  Immunostaining will be reported as mean fluorescence intensity and percentage of cells stained

CONTACTS AND LOCATIONS:
Overall Officials: Hitasha Rupani, BM PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- NIHR Clinical Research Facility, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Researchers and collaborators outside of the study team can submit a request to the PI to access study data at the end of the study for any ethical approved research or external collaborations.